CLINICAL TRIAL: NCT02051452
Title: Reversal of General Anesthesia With Intravenous Methylphenidate
Brief Title: Reversal of General Anesthesia With Methylphenidate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ken Solt, Associate Professor of Anesthesia, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2013P001114
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Post Operative Cognitive Dysfunction; Emergence From Anesthesia
MeSH Terms: interventions — Methylphenidate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Experimental): Methylphenidate
  Interventions: Drug: Methylphenidate
- placebo (Placebo Comparator): Saline
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Methylphenidate
  Other Names: ritalin
  Arms: Methylphenidate
Other: Saline
  Arms: placebo

SUMMARY:
The aim of this study is to investigate whether methylphenidate (Ritalin) can actively induce emergence from general anesthesia in patients having a pancreaticoduodenectomy (Whipple procedure), a pancreatectomy, or a prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* American Society of Anesthesiologists classification 1 or 2
* Scheduled to undergo a pancreaticoduodenectomy or distal pancreatectomy at Massachusetts General Hospital

Exclusion Criteria:

* American Society of Anesthesiologists physical status classification of 3 or beyond.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylphenidate: Patients will receive IV methylphenidate following general anesthesia
- Placebo: Patients will receive IV saline following general anesthesia
Period: Overall Study
Arm/Group | Methylphenidate | Placebo
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 16 MPH patients and 16 placebo patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 7 | 18
  >=65 years | 5 | 9 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Recorded as a measure of safety and tolerability
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

2. Secondary Outcome: Time to Emergence From General Anesthesia
Description: Measured as the time from drug (MPH or saline placebo) administration to extubation
Time Frame: 1-4 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 16 | 16
minutes | 7.5 (3.06) | 8.73 (3.5)

3. Other Pre Specified Outcome: Post Operative Cognitive Function at ½ Hour, 1 Hour and 2 Hours After Emergence as Measured by the Mini Mental Status Exam.
Description: Return to baseline Mini Mental Status Exam (MMSE) score after general anesthesia, measured at 30, 60, and 120 minutes following extubation. Testing is discontinued when the patient returns to their baseline pre-surgery MMSE score. A faster return to baseline represents a better outcome.
Time Frame: up to 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 16 | 16
Participants
  Return to baseline after 30 min | 11 | 8
  Return to baseline after 60 min | 4 | 5
  Return to baseline after 120 min | 1 | 3

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Methylphenidate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT02051452/Prot_SAP_000.pdf